CLINICAL TRIAL: NCT05340582
Title: Co-administration of Acetaminophen With Ibuprofen to Improve Duct-Related Outcomes in Extremely Premature Infants - The ACEDUCT Trial
Brief Title: Co-administration of Acetaminophen With Ibuprofen to Improve Duct-Related Outcomes in Extremely Premature Infants
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); McMaster Children's Hospital (Other); The Rotunda Hospital (Other); John Hunter Hospital (Other Government); Royal Alexandra Hospital (Other); Centre Hospitalier de l'Universite Laval (CHUL) (Unknown); Royal North Shore Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTO 1875
Record Dates: First submitted 2022-03-16; First posted 2022-04-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
Keywords: Preterm Neonates; Patent Ductus Arteriosus; Echocardiography; Acetaminophen; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen; Suspensions; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, double-blinded, placebo controlled, parallel, two-armed, superiority randomized trial comparing two treatment regimens for the first treatment course of PDA in ELGANs
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy (Experimental): Intravenous or enteral ibuprofen, as decided by clinical team, in the standard clinical dose used in participating NICUs (typically, for neonates < 7 days old - 10 mg/kg/dose on day 1, 5 mg/kg/dose q24h on days 2 and 3; for neonates > 7 days old - 20 mg/kg/dose on day 1, 10 mg/kg/dose q24h on days 2 and 3) And study drug (intravenous acetaminophen 15 mg/kg/dose IV q6h for 3 days).
  Interventions: Drug: Acetaminophen Injection; Drug: Ibuprofen 20 mg/mL oral suspension or Ibuprofen lysine 10 mg/mL injection solution (Neoprofen)
- Standard Clinical Practice - Monotherapy (Placebo Comparator): Intravenous or enteral ibuprofen, as decided by clinical team, in the standard clinical dose used in participating NICUs (typically, for neonates < 7 days old - 10 mg/kg/dose on day 1, 5 mg/kg/dose q24h on days 2 and 3; for neonates > 7 days old - 20 mg/kg/dose on day 1, 10 mg/kg/dose q24h on days 2 and 3) And Placebo [(0.9% saline IV q6h for 3 days).
  Interventions: Drug: Ibuprofen 20 mg/mL oral suspension or Ibuprofen lysine 10 mg/mL injection solution (Neoprofen); Other: Sodium chloride 0.9% injection

INTERVENTIONS:
Drug: Acetaminophen Injection — Acetaminophen injection solution 1000 mg/100 mL (10 mg/mL) latex-free plastic bag - dosage for this protocol is 15mg/kg/dose IV four times a day for 3 days
  Arms: Combination Therapy
Drug: Ibuprofen 20 mg/mL oral suspension or Ibuprofen lysine 10 mg/mL injection solution (Neoprofen) — Ibuprofen is not a study drug - standard of care in participating NICUs in the standard clinical dose for neonates (typically, for neonates < 7 days old - 10 mg/kg/dose on day 1, 5 mg/kg/dose q24h on days 2 and 3; for neonates > 7 days old - 20 mg/kg/dose on day 1, 10 mg/kg/dose q24h on days 2 and 3)
Other: Sodium chloride 0.9% injection — Placebo- IV q6h for 3 days
  Arms: Standard Clinical Practice - Monotherapy

SUMMARY:
Patent ductus arteriosus (PDA), the most common cardiovascular complication of prematurity, is associated with higher mortality and morbidities in extremely low gestational age neonates (ELGANs, < 27+0 weeks). Ibuprofen and acetaminophen, which act by reducing prostaglandin synthesis, are the most commonly used first and second line agents for PDA treatment across Canada. However, initial treatment failure with monotherapy is a major problem, occurring in >60% ELGANs. Treatment failure is associated with worsening rates of mortality and bronchopulmonary dysplasia (BPD), while early treatment success can achieve rates comparable to neonates without PDA. Treatment failure resulting in prolonged disease exposure is thought to be a major contributor. Recently, combination therapy with acetaminophen and ibuprofen has emerged as a new treatment regime. Acetaminophen exerts anti-prostaglandin effect through a different receptor site than ibuprofen, providing a biological rationale for their synergistic action.

The objective of this study is to evaluate the clinical impact, efficacy and safety of combination regime (Ibuprofen + IV Acetaminophen) for the first treatment course for PDA in ELGANs vs. Ibuprofen alone (current standard treatment).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <27+0 weeks gestational age
* Permission given by the attending clinician to approach and then consent obtained from parents
* Diagnosis of PDA ≥ 1.5 mm on echocardiography with unrestrictive predominantly left to right shunt
* Designated to receive first treatment course with intravenous or enteral ibuprofen, as decided by the attending team.

Exclusion Criteria:

* Chromosomal anomaly
* Pre-treatment renal dysfunction defined as urine output < 1ml/kg/hour for the previous 24 hours or serum creatinine > 100 micromol/L
* Pre-treatment hepatic dysfunction defined as serum aminotransferase (ALT) > 100 units/L94
* Platelet count <50,000 per microliter
* Permission denied by the attending clinician to approach parents
* Parental consent not available
* Previous exposure to PDA medical treatment with any drug (prophylactic indomethacin use for prevention of intraventricular hemorrhage will not be considered as PDA treatment).

Max Age: 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Composite of pre-discharge mortality or any grade BPD | 36 weeks PMA
  Need for oxygen or positive pressure respiratory support at 36 weeks postmenstrual age (PMA)

SECONDARY OUTCOMES:
PDA treatment success | 6-10 days post treatment initiation
  Defined as PDA closure or becoming insignificant [diameter <1.5 mm]
Renal or hepatic dysfunction | Occurring within 7 days of treatment initiation
  Renal dysfunction defined as urine output < 1ml/kg/hour for the previous 24 hours or serum creatinine > 100 micromol/L; hepatic dysfunction defined as serum aminotransferase (ALT) > 100 units/L
Further exposure to pharmacological PDA treatments | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  As per units' standard practice (not part of study procedures)
Procedure for PDA closure | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  Surgical closure for PDA
Mortality | From date of randomization until date of death (assessed up to a maximum of 250 days after randomization)
  Death during initial tertiary NICU stay
Severity of BPD at 36 weeks PDM using Jensen's criteria | At 36 weeks PDM
  Grade 1, nasal cannula ≤2 L/min; grade 2, nasal cannula >2 L/min or noninvasive positive airway pressure; grade 3, invasive mechanical ventilation
NEC ≥ stage 2A | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  NEC ≥ stage 2A during NICU stay
Duration (days) of invasive or non-invasive respiratory support | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  Days of invasive or non invasive support during NICU say
Need for diuretic use | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  Diuretic use for BPD treatment
Need for systemic steroids | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  Use for BPD treatment
Sepsis | From date of randomization until death, discharge home or discharge to a community hospital (whichever comes first) assessed up to a maximum of 250 days after randomization
  Diagnosis of sepsis during NICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Amish Jain, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (9):
- Australia (2):
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université Laval, Québec, Quebec
- Prince of Wales Hospital, Shatin, NT, Hong Kong
- The Rotunda Hospital, Dublin, Ireland